CLINICAL TRIAL: NCT00735904
Title: Phase 2 Trial Of AG-013736 As First-Line Treatment For Patients With Squamous Non-Small Cell Lung Cancer Receiving Treatment With Cisplatin And Gemcitabine
Brief Title: Trial Of AG-013736, Cisplatin, And Gemcitabine For Patients With Squamous Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061038
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung (NSCLC)
Keywords: AG-013736; axitinib; cisplatin; gemcitabine; NSCLC; squamous cell; lung cancer
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Axitinib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AG-013736/Cisplatin/Gemcitabine (Experimental)
  Interventions: Drug: AG-013736; Drug: gemcitabine; Drug: cisplatin

INTERVENTIONS:
Drug: AG-013736 — AG-013736 5 mg tablets orally, twice daily, until disease progression
  Other Names: axitinib
Drug: gemcitabine — 200-mg or 1 g lyophilized powder, to be administered as 1250 mg/m^2 IV infusion on Day 1 and Day 8 of 21-day cycle. For a maximum of 6 cycles
Drug: cisplatin — 1mg/ml solution or as lyophilized powder, to be administered as 80 mg/m^2 IV infusion on Day 1 of 21-day cycle. For a maximum of 6 cycles

SUMMARY:
This study will evaluate whether AG-013736 when combined with cisplatin and gemcitabine shows activity and is safe in patients with squamous type of non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of squamous NSCLC Stage IIIB with malignant effusion (fluid cytology demonstrating malignant cells required), Stage IV, or recurrent disease after definitive local therapy
* Candidate for primary treatment with cisplatin and gemcitabine
* Presence of measurable disease by RECIST
* Adequate organ function as defined by the following criteria: ECOG performance status of 0 or 1

Exclusion Criteria:

* Prior systemic treatment for Stage IIIB (with malignant effusion) or Stage IV NSCLC.
* One or more lung lesions with cavitation, or any lesion invading or abutting a major blood vessel as assessed by CT or MRI.
* History of hemoptysis > ½ tsp (2.5 ml) of blood per day for a day or more within 1 week of study treatment, or Grade 3 or 4 hemoptysis within 4 weeks of study treatment
* NCI CTCAE Grade 3 hemorrhage from any cause within 4 weeks of study treatment
* Preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart.
* Untreated brain metastases.
* Need for therapeutic anticoagulation, regular use of aspirin (> 325 mg/day), NSAID or other medications known to inhibit platelet function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-12; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Poland (2):
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Wodzislaw Sl.
- Romania (3):
  - Pfizer Investigational Site, Cluj-Napoca, Cluj
  - Pfizer Investigational Site, Bucharest
  - Pfizer Investigational Site, Oradea
- Pfizer Investigational Site, Parktown, South Africa
- Ukraine (4):
  - Pfizer Investigational Site, Dnipropetrovsk
  - Pfizer Investigational Site, Donetsk
  - Pfizer Investigational Site, Kyiv
  - Pfizer Investigational Site, Lviv

REFERENCES:
- [Derived] Bondarenko IM, Ingrosso A, Bycott P, Kim S, Cebotaru CL. Phase II study of axitinib with doublet chemotherapy in patients with advanced squamous non-small-cell lung cancer. BMC Cancer. 2015 May 1;15:339. doi: 10.1186/s12885-015-1350-6. PMID 25929582
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061038&StudyName=Trial%20Of%20AG-013736%2C%20Cisplatin%2C%20And%20Gemcitabine%20For%20Patients%20With%20Squamous%20Non-Small%20Cell%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib + Cisplatin + Gemcitabine: Axitinib (AG-013736) tablet 5 milligram (mg) starting dose orally twice daily continuously along with cisplatin 80 mg per square meter (mg/m^2) intravenous 2 hours infusion on day 1 of each cycle and gemcitabine 1250 mg/m^2 intravenous 30 minutes infusion on days 1 and 8 of each cycle up to 6 cycles (cycle length 21 days), in chemotherapy phase. Axitinib (AG-013736) tablet 5 mg orally twice daily continuously up to 15 cycles (cycle length 28 days), in single agent phase.
Period: Overall Study
Arm/Group | Axitinib + Cisplatin + Gemcitabine
Started | 38
Completed | 0
Not Completed | 38
Not completed — Adverse Event | 3
Not completed — Death | 20
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Study Terminated by Sponsor | 5
Not completed — Other | 8

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib + Cisplatin + Gemcitabine
Number analyzed (Participants) | 38
Age Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed response are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are those with disappearance of all target lesions. PR are those with at least 30 percent decrease in sum of the longest dimensions of target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline until disease progression or discontinuation from the study due to any cause, assessed every 6 weeks during chemotherapy phase and every 8 weeks during single agent phase up to final study visit (Week 78)
Population: Intent-to-treat (ITT) population included all enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib + Cisplatin + Gemcitabine
Number analyzed (Participants) | 38
Percentage of participants | 39.5 [24.0 to 56.6]

2. Secondary Outcome: Overall Survival (OS)
Description: Time in months from the start of study treatment to date of death due to any cause. OS was calculated as (the death date minus the date of first dose of study medication plus 1) divided by 30.4. Death was determined from adverse event data (where outcome was death) or from follow-up contact data (where the participant current status was death).
Time Frame: Baseline until death or assessed every 2 months (up to 28 days after the last dose)
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + Cisplatin + Gemcitabine
Number analyzed (Participants) | 38
Months | 14.2 [11.8 to 23.1]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Time in months from start of study treatment to the first documentation of objective tumor progression or to death due to any cause. PFS calculated as (Months) = (first event date minus first dose date plus 1) divided by 30.4. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline, assessed every 2 months (up to 28 days after the last dose)
Population: ITT population included all enrolled participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + Cisplatin + Gemcitabine
Number analyzed (Participants) | 38
Months | 6.2 [4.5 to 9.3]

4. Secondary Outcome: Duration of Response (DR)
Description: Time in months from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1) divided by 30.4. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 1
Population: DR was calculated for the subgroup of participants from the ITT set, with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Axitinib + Cisplatin + Gemcitabine
Number analyzed (Participants) | 15
Months | 5.78 [4.7 to 7.2]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib + Cisplatin + Gemcitabine
Serious Adverse Events (participants affected / at risk) | 15/38
Other Adverse Events (participants affected / at risk) | 34/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Cisplatin + Gemcitabine (N=38)
Anaemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 2
Fatigue (General disorders) | 1
Multi-organ failure (General disorders) | 1
Lung abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary artery thrombosis (Nervous system disorders) | 1
Pulmonary embolism (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib + Cisplatin + Gemcitabine (N=38)
Anaemia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 6
Chest pain (General disorders) | 4
Fatigue (General disorders) | 6
Hyperthermia (General disorders) | 2
Pyrexia (General disorders) | 2
Influenza (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Creatinine renal clearance decreased (Investigations) | 5
Weight decreased (Investigations) | 9
Decreased appetite (Metabolism and nutrition disorders) | 8
Hemiparesis (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2
Nephropathy toxic (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.